CLINICAL TRIAL: NCT06775821
Title: Epidemiology of Abdominal Aortic Aneurysm With Concomitant Primary Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Kunming Medical University (Other)
Collaborators: The Third Affiliated Hospital of Kunming Medical University (Unknown); Kunming Medical University (Other)
Responsible Party: Principal Investigator, Dr. Kai-Xiong QING, Associate Professor, First Affiliated Hospital of Kunming Medical University
Other Study IDs: CALUNGAAA
Record Dates: First submitted 2024-05-19; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Abdominal Aortic Aneurysm; Primary Lung Cancer; Prevalence
Keywords: Abdominal Aortic Aneurysm; primary lung cancer; epidemiological studies; prevalence
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Fresh AAA samples, fresh Ca lung samples, with organ donors normal aorta and lung tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary lung cancer with concomitant abdominal aortic aneurysm
  Interventions: Device: Ultrasound or CT of the abdominal aorta

INTERVENTIONS:
Device: Ultrasound or CT of the abdominal aorta — Patient underwent ultrasound or CT of the abdominal aorta

SUMMARY:
Retrospective clinical case studies in recent years have shown that most cases of lung cancer and abdominal aortic aneurysm (AAA) are detected at the same time and that there is a wide variation in the prevalence of AAA in patients with primary lung cancer reported in the literature, with some papers suggesting as high as 11%, suggesting that there may be a relationship between the prevalence of the two diseases. However, its exact incidence and mechanism are unknown. Accurate prevention of AAA in patients with primary lung cancer requires more in-depth studies. To solve the above problems, a multi-center prospective epidemiological investigation and mechanism study on the association of AAA in primary lung cancer combined has become particularly urgent. The results of the study will be of great significance for the follow-up treatment and prognosis of lung cancer patients as well as the improvement of long-term survival rate of lung cancer patients, and will also provide scientific basis and clinical guidance for the screening and prevention of AAA in lung cancer patients.

DETAILED DESCRIPTION:
1. research purpose： This study collected detailed basic information, lifestyle habits, past medical history, and laboratory indicators from 2000-3000 outpatient patients with primary lung cancer for data analysis and long-term follow-up. The study analyzed the related factors of lung cancer complicated with AAA, providing direct scientific evidence to better guide lung cancer patients in screening for AAA, identifying common high-risk factors for lung cancer patients complicated with AAA, providing clinical guidance for the prevention of AAA, and reducing the risk of AAA rupture. The research results are of great significance for the subsequent treatment and prognosis of lung cancer patients, as well as improving the long-term survival rate of lung cancer patients. They will also provide scientific basis and clinical guidance for the screening and prevention of AAA in lung cancer patients. Early detection and treatment of AAA can reduce the risk of AAA rupture, greatly improve the prognosis of lung cancer patients with AAA, and enhance their quality of life.
2. research population： The research subjects are patients diagnosed with primary lung cancer at the Third Affiliated Hospital of Kunming Medical University and the First Affiliated Hospital of Kunming Medical University from 1st October 2022 to 30 st April 2025. The expected sample size is about 2000 people, and the age of patients is 20-90 years old. Collect detailed epidemiological data and long-term follow-up data, conduct statistical analysis, and conduct epidemiological investigations.
3. Epidemiological data collection:

3.1 Basic Information: name, gender, ethnicity, age, height, weight, hometown, occupation, education level, ID card, phone number, and medical record number.

3.2 Behavioral Life Information：Whether smoking, smoking index, alcohol consumption, alcohol content and quantity consumed, history of exposure to asbestos products, dietary habits, and history of dust exposure.

3.3 Past medical history and family genetic history: Presence of hypertension, degree of hypertension, blood pressure control medications, and blood pressure control; diabetes mellitus, blood glucose control medications, and blood glucose control; hyperlipidemia, elevated lipid composition, lipid control medications, and lipid control; urologic disorders; family history of vascular disorders; and family history of oncologic disorders.

3.4 Laboratory information: Blood pressure, fasting blood glucose, glycosylated hemoglobin Total cholesterol (TC), triglyceride (TG), high-density lipoprotein-cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C).

3.5 Follow-up information:

1. Information related to primary lung cancer: types of lung tumors (squamous cell carcinoma, adenocarcinoma, small cell/neuroendocrine/other); Staging of lung tumors (stages I, II, III, IV); CNM staging; Differentiation results of lung tumors; Immunohistochemical staining results; Tumor markers (outliers); Tumor genes (outliers); The treatment methods for lung tumors (surgery, radiotherapy, chemotherapy, molecular targeting, immunity, biological therapy, neoadjuvant chemotherapy); Surgical time and bleeding volume.
2. Information related to abdominal aortic aneurysm: whether it is complicated with abdominal aortic aneurysm; Is there a concomitant iliac artery aneurysm; Whether to undergo surgical treatment; Surgical treatment methods (endovascular repair of abdominal aortic aneurysm, open surgery); Surgical time and bleeding volume.
3. Patient prognosis: last follow-up time, time of lung tumor recurrence, whether death occurred, and cause of death.

4.Data entry and analysis At the Department of Thoracic Surgery of the First Affiliated Hospital of Kunming Medical University and the Department of Thoracic Surgery of the Third Affiliated Hospital of Kunming Medical University, patient basic information, laboratory tests, and treatment plans are obtained and filled out from the hospital's medical record system. Epidemiological survey questions are collected at the patient's bedside using a question and answer format to ensure the accuracy and reliability of the epidemiological survey information. All collected data is organized and encoded using REDCap（ https://www.wcrcnet.cn/redcap/ ）Perform data entry. IBM SPSS Statistics 22 will be used to analyze the entered data and identify the risk factors for primary lung cancer combined with AAA.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary lung cancer through clinical or pathological examination

Exclusion Criteria:

* Patients diagnosed with primary lung cancer who refuse to undergo abdominal aortic imaging screening.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The selected subjects for the study were all patients diagnosed with primary lung cancer at the First Affiliated Hospital of Kunming Medical University and the Third Affiliated Hospital of Kunming Medical University from 1st October 2022 to 30 st April 2025, with an estimated sample size of about 2000 people. Detailed epidemiological data and long-term follow-up data were collected and analyzed, and epidemiological investigations were conducted.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of abdominal aortic aneurysm in patients with primary lung cancer | 2022-10-01 to 2025-04-30
  Incidence of abdominal aortic aneurysm in patients with primary lung cancer

SECONDARY OUTCOMES:
Epidemiological analysis | 2022-10-01 to 2025-04-30
  Common pathogenic factors of primary lung cancer with concomitant abdominal aortic aneurysm

CONTACTS AND LOCATIONS:
Overall Officials: Xu-Dong Xiang, MPhil, Study Director — The Third Affiliated Hospital of Kunming Medical University; Ding-yun You, Ph.D., Study Director — Kunming Medical University; Yun-fei Shi, MPhil, Study Director — First Affiliated Hospital of Kunming Medical University; Gui-ming Liu, MBBS, Principal Investigator — The Third Affiliated Hospital of Kunming Medical University; Qing-yan Ma, MBBS, Principal Investigator — Kunming Medical University; Qian Zhu, MBBS, Principal Investigator — The Third Affiliated Hospital of Kunming Medical University; Kai-xiong Qing, ph.D., Study Chair — The Third Affiliated Hospital of Kunming Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The Third Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided
If necessary, upload to make individual participant data (IPD) available to other researchers after the research is completed

REFERENCES:
- [Background] Sakalihasan N, Michel JB, Katsargyris A, Kuivaniemi H, Defraigne JO, Nchimi A, Powell JT, Yoshimura K, Hultgren R. Abdominal aortic aneurysms. Nat Rev Dis Primers. 2018 Oct 18;4(1):34. doi: 10.1038/s41572-018-0030-7. PMID 30337540
- [Background] Schanzer A, Oderich GS. Management of Abdominal Aortic Aneurysms. N Engl J Med. 2021 Oct 28;385(18):1690-1698. doi: 10.1056/NEJMcp2108504. No abstract available. PMID 34706173
- [Background] Golledge J. Abdominal aortic aneurysm: update on pathogenesis and medical treatments. Nat Rev Cardiol. 2019 Apr;16(4):225-242. doi: 10.1038/s41569-018-0114-9. PMID 30443031
- [Result] Alnahhal KI, Urhiafe V, Narayanan M, Irshad A, Salehi P. Prevalence of abdominal aortic aneurysms in patients with lung cancer. J Vasc Surg. 2022 May;75(5):1577-1582.e1. doi: 10.1016/j.jvs.2021.09.037. Epub 2021 Oct 8. PMID 34634421
- [Result] Wiles B, Comito M, Labropoulos N, Santore LA, Bilfinger T. High prevalence of abdominal aortic aneurysms in patients with lung cancer. J Vasc Surg. 2021 Mar;73(3):850-855. doi: 10.1016/j.jvs.2020.05.069. Epub 2020 Jul 2. PMID 32623102
- [Result] Cho HJ, Yoo JH, Kim MH, Ko KJ, Jun KW, Han KD, Hwang JK. Risk of various cancers in adults with abdominal aortic aneurysms. J Vasc Surg. 2023 Jan;77(1):80-88.e2. doi: 10.1016/j.jvs.2022.03.896. Epub 2022 Jul 15. PMID 35850163
- [Result] Hohneck A, Shchetynska-Marinova T, Ruemenapf G, Pancheva M, Hofheinz R, Boda-Heggemann J, Sperk E, Riffel P, Michels J, Borggrefe M, Akin I, Sigl M. Coprevalence and Incidence of Lung Cancer in Patients Screened for Abdominal Aortic Aneurysm. Anticancer Res. 2020 Jul;40(7):4137-4145. doi: 10.21873/anticanres.14413. PMID 32620663
- [Result] Harthun NL, Lau CL. The incidence of pulmonary neoplasms discovered by serial computed tomography scanning after endovascular abdominal aortic aneurysm repair. J Vasc Surg. 2011 Mar;53(3):738-41. doi: 10.1016/j.jvs.2010.09.066. Epub 2010 Dec 3. PMID 21129909
- [Result] Lederlin M, Tredaniel J, Priollet P. [Why screen for lung cancer in patients with arterial disease?]. J Mal Vasc. 2015 Dec;40(6):359-64. doi: 10.1016/j.jmv.2015.07.001. Epub 2015 Aug 12. French. PMID 26276562
- [Result] Erbel R, Aboyans V, Boileau C, Bossone E, Bartolomeo RD, Eggebrecht H, Evangelista A, Falk V, Frank H, Gaemperli O, Grabenwoger M, Haverich A, Iung B, Manolis AJ, Meijboom F, Nienaber CA, Roffi M, Rousseau H, Sechtem U, Sirnes PA, Allmen RS, Vrints CJ; ESC Committee for Practice Guidelines. 2014 ESC Guidelines on the diagnosis and treatment of aortic diseases: Document covering acute and chronic aortic diseases of the thoracic and abdominal aorta of the adult. The Task Force for the Diagnosis and Treatment of Aortic Diseases of the European Society of Cardiology (ESC). Eur Heart J. 2014 Nov 1;35(41):2873-926. doi: 10.1093/eurheartj/ehu281. Epub 2014 Aug 29. No abstract available. PMID 25173340
- [Result] Scorza R, Ghilardi G, De Monti M, Sgroi G. [Current knowledge and unresolved problems in the pathogenesis of abdominal aortic aneurysm]. Minerva Cardioangiol. 1994 Sep;42(9):417-27. Italian. PMID 7991161

DOCUMENTS (1):
  • Informed Consent Form (2025-01-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT06775821/ICF_000.pdf